CLINICAL TRIAL: NCT04885023
Title: Effects of Hippotherapy on Postural Asymmetries and Balance in Adolescents With Idiopathic Scoliosis: a Randomized Controlled Study
Brief Title: Efficacy Hippotherapy on Postural Asymmetries and Balance in Adolescents With Idiopathic Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Batterjee Medical College (Other)
Collaborators: Taif University (Other)
Responsible Party: Principal Investigator, Osama Ragaa Abdelraouf Ibrahim, Professor, Batterjee Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Batterjee Medical College; (TURSP-2020/82) (Other Grant/Funding Number: Taif University, Saudi Arabia)
Record Dates: First submitted 2021-05-04; First posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Idiopathic Scoliosis; Equine-assisted Therapy
Keywords: Hipptherapy; Formateric; Balance; Schroth exercises
MeSH Terms: interventions — Equine-Assisted Therapy

STUDY DESIGN:
Intervention Model Description: A total of 52 patients (15 males and 37 females) participated in the current study, assigned to 2 groups, which were the group A who received hippotherapy combined with Schroth exercises and group B who received only Schroth exercises
Who Masked: Participant, Outcomes Assessor
Masking Description: All participants in two groups in addition to the formetric measurements and Biodex body balance assessors were not aware of the purpose of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Twenty six patients who received hippotherapy combined with Schroth exercises for ten weeks
  Interventions: Other: Hippotherapy
- Control group (Other): Twenty six patients who received only Schroth exercises for ten weeks
  Interventions: Other: Hippotherapy

INTERVENTIONS:
Other: Hippotherapy — The hippotherapy program for 10 weeks
  Other Names: Schroth exercises

SUMMARY:
This study showed that the addition of hippotherapy to Schroth exercises is more effective in improving postural asymmetry and balance ability in adolescents with idiopathic scoliosis compared to Schroth exercises alone. Therefore, this combination should be considered during designing a rehabilitation program for AIS

DETAILED DESCRIPTION:
The hippotherapy program started with a physical therapy assessment to develop specific corrective movements to be practiced while riding the horse based on the direction of the spinal curvature. Interventions were performed by a licensed physical therapist experienced with hippotherapy at two local therapeutic riding centers. The participants received 15 sessions split into two phases over 10 weeks. In the first phase, during the first 5 weeks, they performed 30 minutes of walking and sitting trot training without a stirrup iron once a week. The frequency was then raised to twice a week for the rest of the treatment program. Before the start of the intervention, two familiarization sessions were given to clarify safety guidelines, riding mistakes, and create a riding rapport with the horse. The individuals wore protective helmets during each hippotherapy session and mounted on a moving horse on walk and/or trot performing different positions, namely forward astride, side sitting, backward astride, sometimes with transitions between positions and often while the horse was moving. To restore normal alignment of the spine, participants were also asked to ride without holding on with their hands to perform self-correction movements. Examples of these movements include raising both arms high to decrease the degree of thoracic kyphosis, bending the upper trunk towards the convex side of the curve, raising the arm on the concave side with scapular adduction to level both shoulders. To correct pelvic obliquity, a small pad was put under the hip on the side of the lumbar convexity. Under the instructions of the physical therapist, a leader pulled the horse reins in front to control the horse gait, gait velocity, and orient the horse in different directions . All these movements activate the patient's neuromuscular and sensory reactions.

Both groups performed Schroth exercises that are patient-specific asymmetric exercises with rotational breathing methods used for three-dimensional correction. For the first 2 weeks, there were five 1-h long individual sessions during which the participants were trained in their home exercise program. This was followed by 1-h weekly visits and paired with their daily home exercises. These exercises aimed to provide and promote enhanced postural control by using asymmetrical standing postural exercises specifically designed to restore body balance and mobility. During ground exercises, aid pads were used to build pressure for costal protrusions and/or trunk asymmetry correction. Postural correction was facilitated by rotational breathing exercises focusing on the concave side of the thorax. During the therapy sessions, postural correction principles of the Schroth process, axial elongation, deflection, de-rotation, facilitation, stabilization, were used.

ELIGIBILITY:
Inclusion Criteria:

* AIS,
* all curve types,
* curves with Cobb angle ranged between 10 and 25 degrees,
* a Risser grade 0 to 5, and
* the ability to attend weekly visits.

Exclusion Criteria:

* Children with any significant history of riding horses,
* with diagnosis other than AIS,
* having other treatment which might affect scoliosis,
* having chronic diseases requiring any drug usage,
* presence of other neurologic, muscular or rheumatic diseases, and
* having non-idiopathic scoliosis.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2021-03-07 (Actual)

PRIMARY OUTCOMES:
Scoliotic angle un degrees | 10 weeks
  Measured by formatric 4-D system
Kyphotic angle in degrees | 10 weeks
  Measured by formatric 4-D system
Pelvic obliquity in degrees | 10 weeks
  Measured by formatric 4-D system
Pelvic torsion in degrees | 10 weeks
  Measured by formatric 4-D system
Vertical spinal rotation in degrees | 10 weeks
  Measured by formatric 4-D system

SECONDARY OUTCOMES:
Overall balance index | 10 weeks
  Measured by Biodex Balance System
Anteroposterior balance index | 10 weeks
  Measured by Biodex Balance System
Mediolateral balance index | 10 weeks
  Measured by Biodex Balance System

CONTACTS AND LOCATIONS:
Overall Officials: Amr A AbdelAziem, Ph.D, Principal Investigator — Tyiaf University, Saudi Arabia
Locations (1):
- Batterjee Medical College, Jeddah, Mecca Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
Data Will Be available only for third parties